CLINICAL TRIAL: NCT04284735
Title: Role of Lysophosphatidic Acid and Autotaxin in Rheumatoid Arthritis-associated Interstitial Lung Disease
Brief Title: Lysophosphatidic Acid / Autotaxin Axis in Rheumatoid Lung Disease
Acronym: LYSLUNG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL19_0930; 2019-A03087-50 (Other: ID-RCB)
Record Dates: First submitted 2020-02-18; First posted 2020-02-26 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Interstitial lung disease; Autotaxin; Lysophosphatidic acid
MeSH Terms: conditions — Arthritis, Rheumatoid; Lung Diseases, Interstitial

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Controls (Other): Patients with RA and without ILD
  Interventions: Other: Quantitative ATX and LPA determination in plasma and sputum
- Cases (Other): Patients with RA and ILD
  Interventions: Other: Quantitative ATX and LPA determination in plasma and sputum

INTERVENTIONS:
Other: Quantitative ATX and LPA determination in plasma and sputum — Determination of ATX and LPA levels in plasma and sputum from RA-ILD patients ("cases") and in plasma and sputum from RA patients without ILD ("controls") after sputum induction using hypertonic saline inhalation

SUMMARY:
Rheumatoid arthritis (RA) is a common chronic systemic autoimmune relapsing disease characterized by joint inflammation. Beside arthritis leading to progressive joint damage and loss of function, RA is also associated to extraarticular inflammatory conditions such as interstitial lung disease (ILD). This one develops in 30% of all RA patients with a median survival expectancy of 3 to 10 years once symptomatic. Unfortunately, there is no medical care recommendation so far as the pathophysiology is unknown. However, ILD share many similarities with idiopathic pulmonary fibrosis (IPF).

Autotaxin (ATX), due to its lysophospholipase activity, produces a bioactive lipid, lysophosphatidic acid (LPA) under inflammation. LPA has pleiotropic actions inducing cell proliferation, survival, motility and differentiation. Increased ATX and LPA levels have been detected in synovial fluid of RA patients and in IPF patients. ATX is also currently the target for a phase 3 clinical trial in IPF.

Given the previous described role of ATX/LPA axis in arthritis and inflammation-induced bone loss in RA and the similarities between RA-ILD and IPF, the investigators hypothesized that ATX/LPA axis may be also an attractive drug target for this pulmonary condition in RA and therefore that ATX and LPA may be increased in sputum from RA patients with ILD in comparison with sputum from RA patients without ILD.

ELIGIBILITY:
Inclusion Criteria:

General inclusion criteria

* Subject aged ≥ 18 and ≤ 70 years
* Patient with RA with ACPA in the state phase, meeting ACR / EULAR 2010 criteria
* For female subjects:

  * Likely to procreate: negative pregnancy test at the inclusion visit and use of an effective method of contraception (hormonal contraceptives, intrauterine devices, vasectomized partner, abstinence) started at least 1 month before inclusion and continued during the entire study.
  * Inability to procreate: menopause (absence of a rule for at least 1 year) or hysterectomy or bilateral oophorectomy or tubal ligation.
* Subject having given written consent to participate in the study
* Subject affiliated to the Social Security scheme or benefiting from an equivalent scheme

Additional inclusion criteria for cases (RA patients with PID):

- PID is defined as damage compatible with the thoracic scanner in thin sections according to international criteria with or without associated clinical signs.

Additional inclusion criteria for control patients (RA patients without symptomatology without PID)

- No functional lung complaints

Exclusion Criteria:

General exclusion criteria

* Vulnerable patient within the meaning of current French legislation (deprived of liberty by judicial or administrative decision, under guardianship or curatorship or under the protection of justice)
* Patient not fluent in French
* Woman breastfeeding or planning a pregnancy for the duration of the study
* Patient in exclusion period after participating in another clinical trial or in the process of participating in another clinical trial involving an experimental product
* Patient with occupational exposure to particles known to be responsible for PID (silica, etc.)
* Patient with an autoimmune disease other than RA or an auto-inflammatory disease

Non-inclusion criteria for cases (RA patients with PID):

- Patient with a history of asthma, COPD or any other pulmonary pathology or pulmonary symptom unrelated to PID

Non-inclusion criteria for control patients (RA patients without PID)

- Patient with a history of asthma, COPD, any other pulmonary pathology, any pulmonary symptom or any pulmonary CT abnormality.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03-03 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
ATX and LPA levels in sputum from RA patients with ILD in comparison with sputum from RA patients without ILD | Month 30
  All the samples will be frozen and ATX and LPA levels will be assessed in the plasma and sputum at the same time, at the end of the recruitment.

SECONDARY OUTCOMES:
Correlation between ATX and LPA levels and severity of RA-ILD estimated by tomodensitometry | Month 24
  Determine the correlation between ATX and LPA levels and the severity of CT scan pulmonary involvement*.
  *Diffuse interstitial lung disease is defined as an attack compatible with the thoracic scanner in thin sections according to international criteria with or without associated clinical signs.

CONTACTS AND LOCATIONS:
Overall Officials: Fabienne COURY-LUCAS, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Lyon Sud, Pierre-Bénite, France